CLINICAL TRIAL: NCT00167102
Title: A Double-Blind, Placebo-Controlled, Randomized, Multi-Center Study to Evaluate The Safety and Therapeutic Efficacy of Intramuscular Administration of Alefacept in Patients With Chronic, Severe Scalp Alopecia Areata
Brief Title: Alefacept in Patients With Severe Scalp Alopecia Areata
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Alopecia Areata Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 0506M70377
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Results first posted 2013-04-09 (Estimated); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Alopecia Areata
Keywords: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — Alefacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alefacept (Experimental)
  Interventions: Drug: Alefacept
- Placebo (Placebo Comparator)
  Interventions: Drug: Alefacept

INTERVENTIONS:
Drug: Alefacept — Study participants will receive weekly IM administration of placebo or 15 mg of alefacept for 12 weeks, to be followed by a 12-week post-treatment period during which the safety, efficacy, and durability of effect in treatment responders will be assessed on weeks 2, 4, 8 and 12.

SUMMARY:
The purpose of this study is to examine prospectively the safety and efficacy of alefacept in the treatment of subjects with severe alopecia areata of the scalp. Common features between psoriasis and alopecia areata, including immunologic and therapeutic aspects, suggest that alefacept, which has been shown to be a safe and statistically significant beneficial therapeutic modality for the treatment of psoriasis, may have therapeutic value in alopecia areata.

DETAILED DESCRIPTION:
Alopecia areata (AA) is an autoimmune condition characterised by a T-cell mediated attack on the hair follicle. The inciting antigenic stimulus is unknown. A dense peribulbar lymphocytic infiltrate and reproducible immunologic abnormalities are hallmark features of the condition. The cellular infiltrate primarily consists of activated T-lymphocytes and antigen-presenting Langerhans cells. T-lymphocytes play a critical role in the pathogenesis of disease. The observance of hair regrowth in those with alopecia areata who are treated with cyclosporine, a known inhibitor of T-cell function, further confirms the central role of the T-lymphocytes in the development of the disease.

Activation of T-cells is initiated by interaction of the T-cell receptor with the antigen/major histocompatibility complex on the antigen-presenting cells. Co-stimulatory interactions occur secondarily, including binding of the T-cell CD2 receptor to the antigen-presenting cell ligand LFA-3 (lymphocyte function-associated antigen-3 CD58). Induction of a molecular signaling cascade with resultant T-cell activation and proliferation ensues. Abrogation of this activation may result in diminished or aborted expression of disease, and thus suggests a potential therapeutic role for alefacept in the treatment of alopecia areata. Alefacept is a bioengineered LFA-3/Immunoglobulin fusion protein that binds to the CD2 T-cell receptor and interferes with the ligation of LFA-3. Binding of the immunoglobulin portion of the fusion protein to the FCy receptor on antigen-presenting cells potentiates apoptosis of CD-2 T-cells to thereby reduce the population of activated T-cells.

Psoriasis is a T-cell mediated disorder that shares many immunologic features with alopecia areata. Accordingly, treatments that are effective in psoriasis often prove to be beneficial in alopecia areata. Anthralin, topical and intralesional steroids and cyclosporine are among several therapeutic agents that have efficacy in both disorders. Based on the impressive therapeutic responses seen in those with psoriasis treated with alefacept, a similarly beneficial outcome is tentatively anticipated with treatment of those with alopecia areata.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must give written informed consent and candidates in the US must authorize the release and use of protected health information (PHI)
* Subjects must be between the ages of 18 and 65 inclusive at the time of informed consent
* Must have a diagnosis of scalp alopecia areata as determined by the study investigator
* Must have 50-95% patchy scalp hair loss due to alopecia areata of at least one year duration
* Must have CD4+ T-lymphocyte counts at or above the lower limit of normal as determined by a local laboratory.

Exclusion Criteria:

* History of systemic or cutaneous malignancy other than treated basal cell carcinomas or 3 or less squamous cell carcinomas.
* Nevi or cutaneous lesions currently undiagnosed but suspicious for malignancy.
* Evidence of immunocompromise.
* Advanced or poorly controlled diabetes.
* Unstable cardiovascular disease.
* Clinically significant medical or psychiatric disease as determined by the investigator.
* History of alcohol or drug abuse within 2 years of assessment for study enrollment.
* Serious local infection (e.g. cellulitis, abscess) or systemic infection (e.g. pneumonia, septicemia) within 3 months prior to the first dose of investigational drug.
* Positive PPD history of incompletely treated or untreated tuberculosis.
* Abnormal T-lymphocyte count, and/or liver function tests.
* If female, serum hemoglobin level greater than 1 unit below accepted limit for normal or otherwise abnormal.
* Male subjects with an abnormal serum hemoglobin.
* Known positivity for hepatitis C antigen or hepatitis B surface antigen.
* Known positivity for HIV antibody.
* Diagnosis of diffuse alopecia areata.
* Coexistent androgenetic alopecia which, in males is Norwood-Hamilton stage VI or greater, or in females, Ludwig stage III.
* Prior treatment with alefacept.
* Treatment with another investigational drug within 4 weeks prior to anticipated first treatment dose.
* Unable to practice effective contraception for the duration of the study.
* Females who are nursing, pregnant or planning to become pregnant while in the study.
* Those who have donated blood within a month of date of screening evaluation.
* Concomitant enrollment in other investigational drug study.
* Unwilling to maintain a consistent hair style and to eschew shaving of scalp hair throughout the course of the study.
* Unable to comply with the protocol.
* Other unspecified reasons that contraindicate enrollment in the study, as determined by the study investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2005-07; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Hordinsky, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Alefacept: Weekly IM administration of alefacept,15 mg, for 12 weeks, followed by a 12-week, posttreatment observation period.
- Placebo: Weekly IM administration of placebo, for 12 weeks, followed by a 12-week, posttreatment observation period.
Period: Overall Study
Arm/Group | Alefacept | Placebo
Started | 23 | 22
Completed | 23 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 23 participants were allocated to alefacept 22 participants were allocated to placebo
Groups:
- Alefacept; Placebo: Weekly IM administration of placebo or 15 mg of alefacept for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Alefacept | Placebo | Total
Number analyzed (Participants) | 23 | 22 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 22 | 45
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (10.3) | 34.2 (11.8) | 36.3 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 14 | 32
  Male | 5 | 8 | 13
Region of Enrollment [Number; unit: participants]
  United States | 23 | 22 | 45

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects Achieving at Least a 50% Reduction in Their Scalp Alopecia Areata Severity Scores (SALT Score) From Baseline Values
Description: Assess the therapeutic efficacy of a 12-week regimen of weekly IM administration of alefacept followed by a 12 week observation period in subjects with chronic severe scalp alopecia
Time Frame: 24 weeks
Measure: Number; unit: percentage of participants
Groups:
- Alefacept: Weekly intramuscular administration of alefacept 15mg for 12 weeks
- Placebo: Weekly intramuscular administration of placebo 15 mg for 12 weeks
Arm/Group | Alefacept | Placebo
Number analyzed (Participants) | 23 | 22
percentage of participants | 8.7 | 13.6

2. Primary Outcome: Number of Adverse Events
Description: Number of any adverse event reported throughout the study, regardless of relation to study drug
Time Frame: 24 weeks
Measure: Number; unit: adverse events
Arm/Group | Alefacept | Placebo
Number analyzed (Participants) | 23 | 22
adverse events | 20 | 20

ADVERSE EVENTS:
Arm/Group | Alefacept | Placebo
Serious Adverse Events (participants affected / at risk) | 1/23 | 2/22
Other Adverse Events (participants affected / at risk) | 20/23 | 9/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alefacept (N=23) | Placebo (N=22)
right elbow arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
vomiting and dehydration (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alefacept (N=23) | Placebo (N=22)
Congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Infection (Infections and infestations) | 4 | 3
Cold (Infections and infestations) | 4 | 2
Headaches (General disorders) | 4 | 3
Nausea (Gastrointestinal disorders) | 2 | 1

LIMITATIONS AND CAVEATS:
This study was limited by the number of patients randomized to receive treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No